CLINICAL TRIAL: NCT00334945
Title: Evaluate the Effect of Growth Hormone (GH) Treatment on Fibroblast Growth Factor 23 (a Known Phosphaturic Agent)
Brief Title: Evaluate the Effect of Growth Hormone (GH) Treatment on Fibroblast Growth Factor 23, a Known Phosphaturic Agent
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Ambika Ashraf, M.D., Principal Investigator, University of Alabama at Birmingham
Other Study IDs: X041104010; X3395n; Genentech X3395n (Other Grant/Funding Number: Genentech)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Growth Disorders
Keywords: Fibroblast Growth Factors; Bone development
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Growth Hormone: Patient ages 3-14 years receiving growth hormone for growth hormone deficiency or short stature
- Healthy Children: Children with normal stature ages 3-18 years.

SUMMARY:
The purpose of this study is to evaluate the effect of growth hormone treatment on phosphorus levels in the body. Phosphorus is an important mineral for bone growth. It is well known that growth hormone treatment improves bone density and bone mineral content. The amount of phosphorus is maintained by the kidneys. Fibroblast Growth Factor 23 has recently been recognized to help kidneys control phosphate levels.

DETAILED DESCRIPTION:
This study will compare Fibroblast Growth Factor 23 levels in children with and without growth hormone deficiency. Children with growth hormone deficiency will have levels taken before starting growth hormone replacement and after it has been initiated.

ELIGIBILITY:
Inclusion Criteria:

* Twenty children with significant short stature < 3rd percentile, ages 3-14 years, and referred to Children's Hospital of Alabama
* Normal healthy volunteer children 3-18 years with normal stature

Exclusion Criteria:

* Patients on medication including GH
* Patients with concomitant hormonal abnormalities
* Patients with disorders of calcium and phosphate metabolism
* Active neoplasms
* Closed epiphysis
* Known bone disorders

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children attending Endocrinology clinics of Children's Hospital of Alabama. Ages are 3-14 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Ashraf, MD, Principal Investigator — University of Alabama at Birmingham